CLINICAL TRIAL: NCT00117780
Title: Comparison of Efficacy and Safety of Insulin Detemir Once or Twice Daily in a Basal-Bolus Regimen With Insulin Aspart in Patients With Type 1 Diabetes
Brief Title: Comparison of Insulin Detemir Given Once or Twice Daily in Type 1 Diabetes
Acronym: ADAPT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN304-1708; 2005-001522-88 (EudraCT Number)
Record Dates: First submitted 2005-06-30; First posted 2005-07-08 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Detemir; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: insulin detemir
Drug: insulin aspart

SUMMARY:
This trial is conducted in Europe. The aim of this research study is to compare the efficacy (reduction in HbA1c and in blood glucose levels) of insulin detemir once daily injection compared to insulin detemir twice daily injection administered as basal insulin for the treatment of type 1 diabetes and to verify the safety of use (number and severity of episodes of hypoglycemia, body weight and side effects).

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes for more than 1 year
* Subject treated by any kind of insulin regimen and whatever the number of injections
* HbA1c = 7.5% and = 10%

Exclusion Criteria:

* Type 2 diabetes
* Treatment by oral anti-diabetic drugs
* Severe medical conditions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Actual)
Dates: Start 2005-06; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Mean HbA1c | after 4 months of insulin detemir treatment

SECONDARY OUTCOMES:
HbA1c
Adverse events
Insulin dose requirements during initial 4 months of treatment and during 3 months extension
Weight
Blood glucose
Hypoglycaemia

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (3):
- Novo Nordisk Investigational Site, Aalst, Belgium
- Novo Nordisk Investigational Site, Lille, France
- Novo Nordisk Investigational Site, Luxembourg, Luxembourg

REFERENCES:
- [Result] Le Floch JP, Levy M, Mosnier-Pudar H, Nobels F, Laroche S, Gonbert S, Eschwege E, Fontaine P; Assessment of Detemir Administration in Progressive Treat-to-Target Trial (ADAPT) Study Group. Comparison of once- versus twice-daily administration of insulin detemir, used with mealtime insulin aspart, in basal-bolus therapy for type 1 diabetes: assessment of detemir administration in a progressive treat-to-target trial (ADAPT). Diabetes Care. 2009 Jan;32(1):32-7. doi: 10.2337/dc08-0332. Epub 2008 Oct 22. PMID 18945928
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com